CLINICAL TRIAL: NCT04295408
Title: Efficacy of Pericapsular Nerve Group Block After Total Hip Arthroplasty Surgery
Brief Title: Pericapsular Nerve Group Block for Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Olfa kaabachi, MD, Professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE-IMKO 103/2019
Record Dates: First submitted 2020-02-23; First posted 2020-03-04 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Hip Arthropathy; Postoperative Pain
Keywords: hip arthoplasty; nerve block; analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Saline Solution; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLACEBO (Placebo Comparator): Pericapsular Nerve Group block with 40 ml saline
  Interventions: Procedure: Pericapsular nerve group block with saline solution
- Pericapsular nerve group block (Experimental): Pericapsular Nerve Group block with 2 mg.kg-1Ropivacaine in 40 ml of saline
  Interventions: Procedure: Pericapsular nerve group block with ropivacaine

INTERVENTIONS:
Procedure: Pericapsular nerve group block with saline solution — A curvilinear low-frequency ultrasound probe (2-5MHz) was initially placed in a transverse plane over the AIIS and then aligned with the pubic ramus by rotating the probe counterclockwise approximately 45 degrees. In this view, the IPE, the iliopsoas muscle and tendon, the femoral artery, and pectineus muscle were observed. A 22-gauge, 100-mm needle was inserted from lateral to medial in an in-plane approach to place the tip in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly. Following negative aspiration, the saline solution was injected in 5-mL increments while observing for adequate fluid spread in this plane.a total volune of 40 ml saline solution was injected.
  Arms: PLACEBO
Procedure: Pericapsular nerve group block with ropivacaine — A curvilinear low-frequency ultrasound probe (2-5MHz) was initially placed in a transverse plane over the AIIS and then aligned with the pubic ramus by rotating the probe counterclockwise approximately 45 degrees. In this view, the IPE, the iliopsoas muscle and tendon, the femoral artery, and pectineus muscle were observed. A 22-gauge, 100-mm needle was inserted from lateral to medial in an in-plane approach to place the tip in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly. Following negative aspiration, local anesthetic was injected in 5-mL increments while observing for adequate fluid spread in this plane. a 2 mg.kg-1Ropivacaine in 40 ml of saline was injected
  Arms: Pericapsular nerve group block

SUMMARY:
Controlling pain after hip replacement surgery improves comfort and partient satisfaction. Pain after hip replacement has traditionally been managed using systemic pain medications including acetaminophen and non-steroidal anti-inflammatory drugs. A recent Cochrane review demonstrated that compared to systemic analgesia alone, peripheral nerve blocks reduce postoperative pain with moderate-quality evidence. Pericapsular Nerve Group block is a new technique allowing local anesthetic diffusion to femoral, obturator and accessory obturator nerves and providing a good analgesic effect for hip fracture surgery. Investigators hypothesized that the PENG block could be an interesting alternative to systemic analgesiscs for pain control after total hip replacement.

DETAILED DESCRIPTION:
The aim of the study was to evaluate the efficacy of the PENG block for intra and postoperative pain control in total hip arthroplasty.

it was a monocentric, randomized, controlled and double blind study. Patients scheduled for primary THA with lateral approach under general anesthesia.

Premedication with IV midazolam 1 to 2 mg on arrival to operating theatre. general anesthesia was conducted using fentanyl, propofol and cisatracurium for induction and isoflurane for maintanance patients were randomized using a random table in two groups:

* PENG Block group (PG) who received 2 mg.kg-1Ropivacaine in 40 ml of saline.
* Placebo group (SG) who received 40 ml of saline.

Postoperative analgesia started before extubation of the patient, with:

* IV paracetamol 1g/6h in Day1 and oral paracetamol 1g/8h for 6 days.
* non steroidal anti inflammatory drugs with IM piroxicam 20 mg on day one (at the end of surgery) and oral diclofenac 50 mg/12h for 3 days.
* Morphine PCA for day 1 (24 H) and oral tramadol 50 mg/12h from day 2 to day 6.

ELIGIBILITY:
Inclusion Criteria:

* primary THA with lateral approach under general anesthesia.

Exclusion Criteria:

* Hip fracture,
* allergy to local anesthetics,
* peripheral neuropathy,
* creatinin clearance inferior to 30ml/min,
* weight inferior to 50 Kg or superior to 100 Kg,
* neurological disorder affecting the lower extremity, significant psychiatric conditions,
* patients receiving corticosteroid therapy,
* chronic consumption of opioids (>2 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | day one
  morphine consumption on mg

SECONDARY OUTCOMES:
intraoperative opioid consumption | Day 0
  total intraoperative fentanyl consumption on microg
Pain score after extubation | up to 30 minutes
  simplified numerical score (SNS) after extubation [0=no pain , 10=worst pain].
postoperative pain score | day one
  simplified numerical score (SNS) [0=no pain , 10=worst pain].
Pain score during seating position | day one
  simplified numerical score (SNS) during seating position [0=no pain , 10=worst pain].

CONTACTS AND LOCATIONS:
Overall Officials: khaireddine Raddaoui, MD, Principal Investigator — Tunis El Manar University
Locations (1):
- Institut Kassab D'Orthopedie, Tunis, Tunisia